CLINICAL TRIAL: NCT06637722
Title: Self-management in Patients With Adrenal Insufficiency.
Status: Active, not recruiting | Type: Observational
Sponsor: Region Stockholm (Other Government)
Responsible Party: Sponsor
Other Study IDs: K0000-9980
Record Dates: First submitted 2024-10-02; First posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-09

CONDITIONS: Adrenal Insufficiency
Keywords: Adrenal insufficiency; self-management
MeSH Terms: conditions — Adrenal Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with adrenal insufficiency and their relatives

SUMMARY:
Background: Cortisol deficiency leads to a wide range of clinical consequences. Substitution with glucocorticoids is necessary and demands knowledge and ability to self-management from the patient.

Methods: Longitudinal questionnaire-based observational study including group education.

Research questions: To find out if education in group, enhances patients´ and relatives' knowledge about adequate dose adjustment of cortisone and increases the feeling of safety and QoL in patients with adrenal insufficiency.

ELIGIBILITY:
Inclusion Criteria:

Adrenal insufficiency or relative to a person with adrenal insufficiency

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with adrenal insufficiency cared for at at the endocrinology department at Karolinska university hospital, Örebro university hospital, university hospital linköping or university hospital of Umeå and their relatives.
Sampling Method: Non-Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2015-09 (Actual); Primary Completion 2020-08 (Actual); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Questionnaire | 6 months
  Rate of participants responding accurately regarding stree-dosing in hypothetical situation of different degrees of physical and psychological stress.

IPD SHARING:
Plan to Share IPD: No